CLINICAL TRIAL: NCT06730542
Title: Zanubrutinib in Combination With Pola-R-CHP and High-dose Methotrexate in Patients With Secondary CNS Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juan P. Alderuccio, MD (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor-Investigator, Juan P. Alderuccio, MD, Associate Professor of Clinical, University of Miami
Organization: University of Miami (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240458
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: CNS Lymphoma
MeSH Terms: interventions — zanubrutinib; Methotrexate; polatuzumab vedotin; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib in combination with Pola-R-CHP and in combination with Methotrexate Group (Experimental): Participants will be in this group for up to 2 years
  Interventions: Drug: Zanubrutinib; Drug: Methotrexate; Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib capsules will be self-administered orally by participants at a starting dose of 160 mg twice a day (BID) or 320 mg once a day (QD)* at the beginning of Cycle 2 of Pola-R-CHP therapy.
Drug: Methotrexate — Participants will receive Methotrexate as per standard of care (SOC).
Drug: Polatuzumab Vedotin — Participants will receive Polatuzumab Vedotin as per standard of care (SOC).
Drug: Rituximab — Participants will receive Rituximab as per standard of care (SOC), as part of combination standard of care Pola-R-CHP therapy.
Drug: Cyclophosphamide — Participants will receive Cyclophosphamide as per standard of care (SOC), as part of combination standard of care Pola-R-CHP therapy.
Drug: Doxorubicin — Participants will receive Doxorubicin as per standard of care (SOC), as part of combination standard of care Pola-R-CHP therapy.
Drug: Prednisone — Participants will receive Prednisone as per standard of care (SOC), as part of combination standard of care Pola-R-CHP therapy.

SUMMARY:
The purpose of this study is to is to determine the effects (good and bad) of Zanubrutinib in Combination with Pola-R-CHP and High-dose Methotrexate in patients with Secondary Central Nervous System (CNS) Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age on the day of signing the informed consent form (or the legal age of consent in the jurisdiction in which the study is taking place).
2. Patients must have histologic confirmation of large B-cell lymphoma (LBCL) defined by the World Health Organization (WHO) classification. All LBCL subtypes are acceptable. Note: Patients with prior treatment for indolent lymphoma are still eligible for participation as long as they did not receive anthracycline-based therapy.
3. Baseline 18-fluorodeoxyglucose (FDG)-positron emission tomography scan/computed tomography (PET/CT) must demonstrate FDG avid lesions compatible with CT-defined anatomical tumor sites (Note: FDG-PET/CT is not mandatory, and patients with CT scans only will be eligible for study entry as well). Patients should have at least 1 measurable site of disease per Lugano classification in FDG-PET/CT or CT scans.
4. Presence of systemic and CNS involvement (brain, cerebellum, brainstem, meninges, cranial nerves, eyes, spinal cord, or a combination of these) at presentation.
5. Determination of CNS involvement can be by brain biopsy, cerebrospinal fluid (CSF) evaluation by cytology and/or flow cytometry, neuroimaging, or strong clinical suspicion by Investigator for which CNS targeted therapy is recommended (ie, numb chin syndrome in patients with high CNS involvement risk).
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2, except due to lymphoma involvement.
7. Life expectancy of greater than ≥ 3 months.
8. Women should avoid becoming pregnant while taking zanubrutinib and for up to 90 days after ending treatment. Therefore, women of childbearing potential must use highly effective contraceptive measures while taking zanubrutininb and for up to 90 days after stopping treatment. It is currently unknown whether zanubrutinib may reduce the effectiveness of hormonal contraceptives, and therefore women using hormonal contraceptives should add a barrier method. Pregnancy testing is recommended for women of reproductive potential prior to initiating therapy.

   Agreement to use contraception during study participation.
   1. Female patients of childbearing potential must use highly effective methods of contraception. Recommended acceptable contraception methods are included in Section 5.12.
   2. Patients using hormonal contraceptives (eg, birth control pills or devices) must use a barrier method of contraception (eg, condoms) as well.
   3. A woman is considered of childbearing potential, ie, fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.
   4. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause.
9. Male patients with a female partner of childbearing potential are eligible if they abstained, are vasectomized or if they agree to the use of barrier contraception with other methods described above during the study treatment period and for 90 days after the last dose of zanubrutinib.
10. Patients must have normal organ and marrow function as defined below:

    1. Absolute neutrophil count (ANC) > 1,000 cells/mm3 independent of growth factor support within 7 days of study entry (≥ 750 cells/mm3 if lymphoma involvement of the bone marrow or spleen).
    2. Platelets ≥ 75,000 platelets/mm3 independent of transfusion support within 7 days of study entry (≥ 50,000/mm3 independent of transfusion support within 7 days of study entry if lymphoma involvement of the bone marrow or spleen).
    3. Hemoglobin > 9 g/dL or > 8 g/dL in case of bone marrow involvement by lymphoma independent of transfusion support within 7 days of study entry.
    4. Serum total bilirubin ≤ 2 x upper limit of normal (ULN; except patients with Gilberts syndrome).
    5. Aspartate aminotransferase (AST; serum glutamic-oxaloacetic transaminase (SGOT)) and alanine transaminase (ALT); serum glutamic-pyruvic transaminase (SGPT)) ≤2.5 x institutional ULN (≤3x institutional ULN if lymphoma involvement of the liver).
    6. Creatinine within normal institutional limits, or creatinine clearance ≥ 40 mL/min (as estimated by the Cockcroft-Gault equation or alternative formula according to institutional guidelines) for patients with creatinine levels above institutional normal.
11. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments (SoA).

Exclusion Criteria:

1. Primary CNS lymphoma without evidence of systemic lymphoma.
2. Prior systemic lymphoma therapy (Note: 1 cycle of an anthracycline based regimen, such as rituximab, cyclophosphamide, hydroxydaunorubicin, oncovin, and prednisone (R-CHOP), polatuzumab vedotin, rituximab, cyclophosphamide, doxorubicin, and prednisone (pola-R-CHP), dose-adjusted etoposide phosphate, prednisone, oncovin, cyclophosphamide, hydroxydaunorubicin, and rituximab (EPOCH-R), or rituximab, cyclophosphamide, vincristine, doxorubicin, and methotrexate (R-Codox-M), and/or 1 dose of intrathecal therapy, will be allowed before enrollment [Section 5.9]). Note: Patients with prior treatment for indolent lymphoma are still eligible for participation as long as they did not receive anthracycline-based therapy.
3. Any uncontrolled or clinically significant cardiovascular disease including the following:

   1. Myocardial infarction within 6 months before screening;
   2. Unstable angina within 3 months before screening;
   3. New York Heart Association class III or IV congestive heart failure;
   4. History of clinically significant arrhythmias (eg, sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes).
   5. Uncontrolled hypertension as indicated by ≥ 2 consecutive blood pressure measurements showing systolic blood pressure > 170 mm Hg and/or diastolic blood pressure > 105 mm Hg at screening.
   6. QT interval corrected with Fridericia's formula (QTcF) > 450 msec or other significant electrocardiogram (EKG) abnormalities, including second-degree atrioventricular block Type II or third-degree atrioventricular block.
4. Active and/or ongoing autoimmune anemia and/or autoimmune thrombocytopenia (eg, idiopathic thrombocytopenia purpura).
5. Uncontrolled intercurrent illness such as liver cirrhosis, autoimmune disorder requiring immunosuppression or long-term corticosteroids (> 10 mg daily prednisone equivalent), or any other serious medical condition, laboratory abnormality, or psychiatric illness which would compromise ability to comply with study procedures.
6. Severe or debilitating pulmonary disease.
7. Concurrent malignancy requiring active therapy.
8. Prior malignancy within the past 3 years, except for curatively treated basal or squamous cell skin cancer, non-muscle-invasive bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancer.
9. Active fungal, bacterial and/or viral infection requiring systemic therapy.
10. Breastfeeding or pregnant women.
11. Known active infection with HIV, or serologic status reflecting active hepatitis B or C infection as follows:

    1. Patients with positive HIV test and undetectable viral load will be eligible for this study.
    2. Presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) DNA is undetectable (< 20 IU), and if they are willing to undergo monitoring every 4 weeks for HBV reactivation.
    3. Presence of hepatitis C virus (HCV) antibody. Patients with presence of HCV antibody are eligible if HCV RNA is undetectable. For more information regarding hepatitis B and C testing, please refer to Section 9.2.5.4.
12. Patients with impaired decision-making capacity.
13. Ongoing treatment with medications that are strong cytochrome P450 (CYP), family 3, subfamily A (CYP3A) inducers.
14. Underlying medical conditions that, in the Investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs.
15. Unable to swallow capsules or disease significantly affecting gastrointestinal function, such as malabsorption syndrome, stomach or small bowel resection, bariatric surgery procedures, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
16. History of severe bleeding disorder, such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention.
17. History of stroke or intracranial hemorrhage within 180 days before the first dose of zanubrutinib.
18. Major surgery within 4 weeks of the first dose of zanubrutinib. Major surgery is defined as open-heart, reconstructive, transplant, removal of a brain tumor or a damaged kidney surgery.
19. The patient requires treatment with warfarin, warfarin derivatives, or other vitamin K antagonists.
20. Vaccination or requirement for vaccination with a live vaccine within 28 days prior to the first dose of study drug or at any time during planned study treatment.
21. Hypersensitivity to zanubrutinib, any components of pola-R-CHP, regimen, and/or high-dose (HD) methotrexate (MTX), or any of the other ingredients of the applicable study medications.
22. Concurrent participation in another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities (DLTs) | Up to 21 days
  The number of participants experiencing dose-limiting toxicities (DLTs) after starting study therapy. Toxicity will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to 5 years
  Overall response rate (ORR) is defined as the proportion of participants with complete response (CR) or partial response (PR) as the best response.
Number of Patients achieving conversion from PR to CR | Up to 5 years
  Conversion from PR to CR will be assessed by the number of patients achieving an initial PR followed by how many will achieve a subsequent CR by Lugano response criteria.
  Partial response (PR) will be calculated by a Deauville score of 4 or 5 with reduced uptake from baseline, and complete response (CR) is defined as a Deauville score of ≤ 3.
Progression-Free Survival (PFS) | Up to 5 years
  Progression-free survival (PFS) is defined as the elapsed time in years from the start of treatment until disease progression or death, whichever is earlier. Participants who remain alive without progression will be censored at the last documented disease assessment date.
Overall Survival (OS) | Up to 5 years
  Overall survival (OS) is defined as the elapsed time in years from the start of treatment until death from any cause. Alive participants will be censored at the last date known to be alive.
Number of participants experiencing treatment-related adverse events (AEs) | Up to 42 months
  The number of participants experiencing treatment-related adverse events (AEs). AEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.
Number of participants experiencing treatment-related serious adverse events (SAEs) | Up to 42 months
  The number of participants experiencing treatment-related serious adverse events (SAEs). SAEs will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, per physician discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Juan P Alderuccio, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No